CLINICAL TRIAL: NCT02572232
Title: Comparison of Three Different Supraglottic Airway Devices and Endotracheal Intubation in Pediatric Difficult Airway Situations in a Manikin
Brief Title: Supraglottic Airway Devices in Pediatric Difficult Airway Situations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Frass, Univ.Prof.Dr., Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1805/2015
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Airway Morbidity; Emergencies
MeSH Terms: conditions — Emergencies | interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combitube, Easytube, Laryngeal masks (Experimental): Combitube, Easytube, Laryngeal mask airway are intubated in pediatric airway manikins by probands in randomized order.
  Interventions: Device: Combitube, Easytube, Laryngeal masks

INTERVENTIONS:
Device: Combitube, Easytube, Laryngeal masks — Supraglottic airway device

SUMMARY:
The purpose of the study is to compare three supraglottic airway devices (Combitube, Easytube, laryngeal mask airway) to endotracheal intubation in a simulated difficult airway scenario in a pediatric manikin.

DETAILED DESCRIPTION:
Supraglottic airway devices (SAD) have been designed for the "cannot intubate, cannot ventilate" scenario in prehospital as well as intrahospital settings and are utilized in medical emergency services and emergency departments all over the world, not only for anticipated and unanticipated difficult airway situations but also as an airway device used by non-anesthesiologists or in situations where only limited practice is possible. Securing an airway in a pediatric emergency situation is crucial. Unfortunately, pediatricians usually lack the required skills and regular practice to perform endotracheal intubation (ETI, which is the gold standard for securing an airway) quickly and safely. SADs would pose a safe and feasible alternative to ETI. However, no studies on this topic are available. The investigators therefore wanted to evaluate three different SADs (Combitube, Easytube, laryngeal mask airway) in simulated difficult airway situations in a pediatric manikin in comparison to ETI.

ELIGIBILITY:
Inclusion Criteria:

* pediatricians
* residents
* interns
* written informed consent form

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Time to successful ventilation | 1 min

SECONDARY OUTCOMES:
Success rate | 1 min
Rating of the device (questionnaire) | 1 min
  questionnaire, ratings from 1 (best) to 5 (worst)
Re-assessment of success rate after 3 months | 3 months
Re-assessment of time to successful ventilation after 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Frass, Prof. Dr., Study Chair — Medical University of Vienna